CLINICAL TRIAL: NCT00314496
Title: Development of MR Simulation for Treatment Planning
Brief Title: Development of Magnetic Resonance (MR) Simulation for Treatment Planning
Status: Completed | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: EX-0004
Record Dates: First submitted 2006-04-11; First posted 2006-04-14 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2012-01

CONDITIONS: Healthy

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Retrospectively have access to MR images of patients to develop software that:

1. segment images
2. convert MR values to electron density and then
3. entered into a dose calculation system

The project involves software development of data that is already available. No intervention is made at this point.

ELIGIBILITY:
Inclusion Criteria:

* Subject 18 years of age and older

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with conform histological diagnosis of glioblastoma multiforme signed the consent forms and were willing to go for curative radiation treatment with temozolomide
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2005-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gino Fallone, PhD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada